CLINICAL TRIAL: NCT03587038
Title: Feasibility Pilot Study of OKN-007 in Combination With Adjuvant Temozolomide Chemoradiotherapy in Patients With Newly Diagnosed Glioblastoma
Brief Title: OKN-007 in Combination With Adjuvant Temozolomide Chemoradiotherapy for Newly Diagnosed Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-Oblato-001; OKN-007 (Other Grant/Funding Number: Oblato Inc)
Record Dates: First submitted 2018-06-04; First posted 2018-07-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — OKN 007; Temozolomide; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OKN-007 3 days per week plus temozolomide (Experimental): OKN-007: 60 mg/kg, IV, 3 times a week Temozolomide: 75 mg/m2, oral, once daily for 42 days Radiotherapy: 60 Gy administered in 30 fractions
  Interventions: Drug: OKN 007; Drug: Temozolomide; Radiation: Photon/Proton IMRT
- OKN-007 5 days per week and temozolomide (Experimental): OKN-007: 60 mg/kg, IV, 5 times a week Temozolomide: 75 mg/m2, oral, once daily for 42 days Radiotherapy: 60 Gy administered in 30 fractions
  Interventions: Drug: OKN 007; Drug: Temozolomide; Radiation: Photon/Proton IMRT

INTERVENTIONS:
Drug: OKN 007 — 400 mg OKN-007/mL in a phosphate buffer
Drug: Temozolomide — 75 mg/m2
Radiation: Photon/Proton IMRT — standard of care treatment to be given 1 to 2 hours after OKN-007

SUMMARY:
This is a pilot study exploring the potential benefit of adding OKN-007 with Temozolomide for treatment in patients with malignant Glioblastoma undergoing adjuvant concomitant radiotherapy. This drug combination is expected to have an anti-cancer effect in patients who have experienced disease progression after first line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients have newly diagnosed histologically proven WHO grade III or grade IV Glioblastoma Multiforme (GBM).
* Patients at initial presentation of GBM must undergo an adequate surgical resection of the primary lesion; patients must be registered within 49 days (7 weeks) of the surgery.
* Patients must have available and be willing to submit a minimum of five unstained slides tumor tissue specimens from the GBM surgery or open biopsy for MGMT status analysis and molecular profile analysis.
* ECOG performance status within 0 - 2
* Full recovery (< grade 1) from the adverse events associated with prior surgery or any earlier intervention and a minimum of 28 days from the administration of any investigational agent
* Adequate renal, liver and bone marrow function: Leukocytes >3,000/mcL; Absolute neutrophil count >1,500/mcL; Platelets >100,000/mcL; AST / ALT (SGPT) <2.5 x ULN; Total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN) (except Gilbert's Syndrome, who must have a total bilirubin < 3.0 mg/dL); Creatinine within normal limits
* Patients must be ≥ 18 years of age
* Patients must be willing to have blood draws for PK analysis
* All patients must have a CT or MRI of the brain within 14 days prior to registration. The brain CT or MRI should be performed with intravenous contrast (unless contraindicated).
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent for this protocol in accordance with institutional and federal guidelines.
* Life expectancy ≥ 3 months, allowing adequate follow up of toxicity evaluation and progression-free survival evaluation;
* Female patient, if of childbearing potential, has a negative serum pregnancy test within 72 hours of taking study medication and agrees to abstain from activities that could result in pregnancy from enrollment through 120 days after the last dose of study treatment
* Male patient agrees to use an adequate method of contraception
* Birth control should be used from the signing of the patient consent form and for 120 days following the last dose of study treatment.
* In addition, men must not donate sperm during study therapy and for 120 days after receiving the last dose of study treatment.

Exclusion Criteria:

* Second primary malignancy (except adequately treated basal cell carcinoma of the skin).
* Patients who had another malignancy in the past, but have been free of active disease for more than 2 years, are eligible
* Have received treatment within the last 28 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Serious concomitant systemic disorders (for example, active infection or abnormal electrocardiogram (ECG) indicative of cardiac disease) that, in the opinion of the investigator, would compromise the safety of the patient and his/her ability to complete the study
* Patients with moderate or severe renal impairment (calculated creatinine clearance of < 60 mL/min)
* Patients with sodium, potassium, or creatinine serum electrolytes > grade 2.
* Screening ECG abnormality documented by the investigator as medically significant
* Inability to comply with protocol or study procedures.
* Women who are pregnant or breastfeeding.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose and the type of dose limiting toxicities | 5 years
  To determine how well patients are able to tolerate combination of OKN-007, temozolomide, and radiotherapy. Adverse events will be tabulated using MedDRA. The severity of the AE will be graded by the Investigator using the NCI CTCAE, version 4.03.

SECONDARY OUTCOMES:
Number of participants who experience progression-free survival | 5 years
  To evaluate the proportion of patients who receive combination OKN-007 and TMZ who do not experience progression
Number of participants who comply with study treatment plan | 5 years
  To evaluate the clinical compliance of participants receiving combination OKN-007 and TMZ
Number of participants who are able to receive a reduction in steroid dose | 5 years
  To evaluate whether study drug combination allows for a reduced steroid dosage
Number of participants who experience overall survival | 5 years
  To evaluate the proportion of patients who receive combination OKN-007 and TMZ who experience overall survival

CONTACTS AND LOCATIONS:
Overall Officials: James Battiste, MD, Principal Investigator — Principal Investigator
Locations (1):
- Stephenson Cancer Center, University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States